CLINICAL TRIAL: NCT04832347
Title: Comparison of the Effectiveness of Exercise and Vagus Therapy in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinop University (Other)
Responsible Party: Principal Investigator, SEFA HAKTAN HATIK, Lecturer, PT, MSc, PhD(c), Sinop University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VNS002
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy; Activity, Motor; Sleep; Stress, Physiological; Fatigue
Keywords: Exercise; Vagus therapy; Autonomic nervous system
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Exercise; Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Experimental): Exercise group will be given stabilization exercises for a total of 24 sessions, 3 times a week for 8 weeks, each session for 45 minutes.
  Interventions: Other: Exercise
- Vagus group (Experimental): Vagus therapy will be applied to Group 2 for 8 weeks, 3 times a week for a total of 24 sessions, each session for 30 minutes.
  Interventions: Other: Vagus Nerve Stimulation
- Control group (No Intervention): Control group will be followed as a control group and no application will be made.

INTERVENTIONS:
Other: Exercise — Exercise Group will be given stabilization exercises for a total of 24 sessions, 3 times a week for 8 weeks, each session for 45 minutes.
  Arms: Exercise group
Other: Vagus Nerve Stimulation — Vagus therapy will be applied for 8 weeks, 3 times a week for a total of 24 sessions, each session for 30 minutes.
  Arms: Vagus group

SUMMARY:
Objective: Sympathetic activity starts to increase during exercise. At the end of the exercise, while sympathetic activation decreases, parasympathetic activity increases. Sympathetic and parasympathetic excursions achieve homeostasis. Most of the parasympathetic activity effects are vagus code. It is aimed to compare the comparison of exercise and vagus therapy in these healthy individuals.

DETAILED DESCRIPTION:
Objective: The aim of this study is to compare the effectiveness of stabilization exercise and vagus nerve stimulation on healthy individuals.

Research Method: This randomized controlled trial; It is planned to be carried out on students and administrative / academic staff at Gümüşhane University.

First of all, the application will be explained to the individuals and online consent will be obtained from the individuals for the application.

Group 1 will be given stabilization exercises. Vagus therapy will be applied to Group 2. Group 3 will be followed as a control group and no application will be made.

Evaluations;

1. Evaluation of autonomous parameters; It was planned to measure pulse and heart rate variability.
2. Chest circumference measurement
3. In addition, it is planned to use "Perceived Stress Scale", "Pitsburg Sleep Quality Scale" and "Fatigue Severity Scale" questionnaires.

All individuals were planned to be evaluated before, after and 1 month after the application.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer individuals (Female and Male),
* Individuals between the ages of 18-50,
* Obtaining the necessary consent for the study,
* No trauma or surgery history in the last 6 months,
* Does not have any chronic disease (Obesity, Diabetes, Hypertension, Osteoporosis)

Exclusion Criteria:

* Individuals not wanting to continue working.
* Individuals having disability during the work process

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-04-30 (Estimated); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-07-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of autonomous parameters | Change from Systolic / diastolic blood pressure (mmHg) at 2 months.
  Systolic / diastolic blood pressure (mmHg) will be measured with the Braun sphygmomanometer.

SECONDARY OUTCOMES:
Chest circumference measurement | Change from a tape measure in the axillary, xiphoid and subcostal regions while at normal (cm) at 2 months, max inspiratory(cm) and max expiration(cm)
  İt was measured with a tape measure in the axillary, xiphoid and subcostal regions while at normal (cm), max inspiratory(cm) and max expiration(cm).
Perceived Stress Scale | Change of the scores obtained in the questionnaires at 2 months.
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress.PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
Pitsburg Sleep Quality Scale | Change of the scores obtained in the questionnaires at 2 months.
  The PSQI was developed by Buysse et al43 in 1989 and is a 24-question instrument. The PSQI provides a quantitative measurement of sleep quality that is used to describe good and bad sleep. The PSQI has 7 subscales: (1) subjective sleep quality (component 1); (2) sleep latency (component 2); (3) sleep duration (component 3); (4) habitual sleep activity (component 4); (5) sleep disturbances (component 5); (6) use of sleep medication (component 6); (7) daytime dysfunction (component 7). A high total score from the instrument reflects poor quality of sleep. The instrument does not indicate whether or not there is a sleep disturbance or how widespread the sleep disturbances are, if present. However, a total PSQI score of ≥ 5 has been determined to be poor sleep quality.
Fatigue Severity Scale | Change of the scores obtained in the questionnaires at 2 months.
  The FSS, which was published in 1989 by Krupp, has nine items. For each question, the patient is asked to choose a number from 1 to 7 that indicates how much the patient agrees with each statement, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Sefa Haktan Hatık, Sinop, Turkeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No